CLINICAL TRIAL: NCT02003872
Title: The Long Term Effect of Adjustable Spaatz 3 Intragastric Balloon on Weight Loss
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopeed due to lack of recruitment
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Alon Lang, Senior physician GI department, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0670-13-SMC
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Obesity; Diabetes; Hypertension
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spattz 3 intragastric balloon (Experimental): obese patients, . BMI ≥ 35 kg/m² or BMI ≥ 30 kg/m² and hypertension or diabetes mellitus. All will have the intragastric balloon
  Interventions: Device: Spatz 3 intragastric balloon

INTERVENTIONS:
Device: Spatz 3 intragastric balloon — Intra gastric balloon implanted using gastroscopy

SUMMARY:
This is an open-label trial investigating the effect of Spatz 3 intragastric balloon on weight loss on obesity and associated co- morbidities.

The study aim is to evaluate the effect of the intra gastric balloon on weight reduction and on related co- morbidities during 1 year of balloon implantation and a year following explantation.

ELIGIBILITY:
Inclusion Criteria:

- 1. Subjects willing to comply with study requirements and have signed an informed consent form.

2. Age 18-70 3. BMI ≥ 35 kg/m² or BMI ≥ 30 kg/m² and hypertension or diabetes mellitus 4. Documented negative pregnancy test in women of childbearing potential. 5. Women of childbearing potential agree to remain on contraceptives for the duration of their trial participation.

Exclusion Criteria:

* 1. Subjects receiving any prescription or over the counter weight loss medication within 30 days prior to randomization (including GLP-1 analogs).

  2. Previous GI surgery that could preclude the ability to place the device. 3. Subjects with a history of abnormal GI anatomical findings documented on imaging study, which in the opinion of the investigator, may impair implantation of the IGB device 4. Subjects with severe GERD that are not responding to Proton Pump Inhibitor (PPI) 5. Known abnormal pathologies or conditions of the upper gastrointestinal tract.

  6. Subjects with symptomatic gallstones within 6 months prior to randomization 7. Coagulopathy defined as hgb <10g/dl and platelet < 100,000/ml or diagnosis of hemophilia, factor X deficiencies or fibrinogen abnormalities 8. Subjects requiring prescription antithrombotic therapy (i.e. anticoagulant or antiplatelet agent) 9. Subjects unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) or any other drugs with bleeding as a potential side effect during the study duration.

  10. Subject is or has been enrolled in another investigational study within 3 months of participation into the current study 11. Subjects not residing within a 3 hour driving distance of the study center.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Excess weight loss | 2 years

SECONDARY OUTCOMES:
liver fat infiltration | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alon Lang, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel